CLINICAL TRIAL: NCT06419335
Title: Reducing Fatigue With CoQ10 Supplementation in Patients With Crohn's Disease Study
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 855592
Record Dates: First submitted 2024-05-07; First posted 2024-05-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease; Healthy
MeSH Terms: conditions — Crohn Disease | interventions — coenzyme Q10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 Crohn's Disease Patients with Fatigue (Experimental)
  Interventions: Drug: CoQ10
- Cohort 2 Crohn's Disease without Fatigue (No Intervention)
- Cohort 3 Healthy Volunteers (Experimental)
  Interventions: Drug: CoQ10

INTERVENTIONS:
Drug: CoQ10 — The core component of this pilot study will be a single center open label randomized trial comparing low dose and high dose CoQ10 among 30 patients with Crohn's disease and fatigue (Cohort 1) and 15 healthy volunteers (Cohort 3).
  Arms: Cohort 1 Crohn's Disease Patients with Fatigue; Cohort 3 Healthy Volunteers

SUMMARY:
This study includes an open label clinical trial comparing two doses of CoQ10 for 8 weeks to improve fatigue among patients with Crohn's disease and a prospective cohort study of healthy controls taking CoQ10 for 2 weeks. Additionally, among 15 participants who do not meet the fatigue threshold for the open label trial, the investigators will measure CoQ10 levels in blood and fasting urine, as well as complete the same data collection.

Hypotheses

1. Fatigue will improve with CoQ10 and there will be a dose response with greater improvement with higher dose as measured by the Patient Reported Outcomes Measurement Information Systems Fatigue PROMIS Fatigue 7a instrument.
2. Fatigue will improve when measured with other fatigue scales in a similar dose dependent manner and that general and physical fatigue will improve more than mental fatigue.
3. CoQ10 will improve quality of life as measured with the short Inflammatory Bowel Disease Questionnaire (sIBDQ).

ELIGIBILITY:
Inclusion Criteria for all study participants

To be eligible for this study all study participants must meet the following:

1. Provide informed consent
2. Male or female, age 18-70
3. Ability to take an oral medication
4. Willingness and ability to do electronic surveys

Additional inclusion criteria for Cohort 1 and Cohort 2 participants:

1. Must have Crohn's disease for at least 3 months
2. Must be on stable medication regimen for Crohn's disease for at least 4 weeks
3. Clinically quiescent Crohn's disease based on the Patient Reported Outcome -Crohn's Disease (PRO2) average score for up to 7 days - daily liquid or very soft stool frequency of ≤1.5 and abdominal pain ≤1.0 5.3 Additional inclusion criteria for Cohort 1

1. Prescreening PROMIS Fatigue 7a T score >60 5.4 Additional inclusion criteria for Cohort 2 and 3

1. Prescreening PROMIS Fatigue 7a T score <55

Exclusion Criteria - for all study participants

1. Pregnant or lactating - a blood pregnancy test will be administered - fatigue is common with pregnancy and the post-partum period and is more likely to be unrelated to Crohn's
2. Chronic fatigue syndrome - noted in the medical record or self-reported
3. Depression as measured with PROMIS Depression scale 7a with T score >=60
4. New York Heart Association (NYHA) class 3 or greater heart failure - if noted in the medical record
5. Untreated sleep apnea
6. Abnormal Thyroid Stimulating Hormone (TSH) - <0.45 μlU/mL or >5.33 μlU/mL
7. Iron deficiency or anemia - ferritin < 20 without anemia or <100 with anemia (hemoglobin < 12g/dL in females or 13.5 g/dL in males) on the screening laboratory tests
8. B12 deficiency - <180 pg/mL on the screening laboratory tests
9. Stage 3B or higher Chronic Kidney Disease (CKD) - based on an estimated glomerular filtration rate (eGFR) < 45 ml/min on the screening laboratory tests
10. Diagnosis of cirrhosis - if noted in the medical record or self-reported
11. Diagnosis of primary sclerosing cholangitis
12. Diagnosis with hepatitis C without evidence of successful eradication
13. Cancer and receiving chemotherapy - if noted in the medical record or self-reported
14. Multiple Sclerosis - self-reported on in chart.
15. Taking systemic corticosteroids (e.g. prednisone or budesonide), not including single doses given to prevent adverse reactions to a medication or contrast agent
16. Taking warfarin - if noted in the medical record or self-reported
17. Diabetes requiring medication - if noted in the medical record or self-reported
18. Symptoms of an infection in the last 2 weeks - self-reported
19. Any other comorbidity or condition that the PI thinks is a contraindication to participation in this study

Exclusion Criteria for Cohorts 1 and 3

1. Previous intolerance to CoQ10

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Assess improved fatigue among patients with Crohn's Disease | 8 weeks
  The primary objective of this study is to assess whether there is sufficient evidence of a change (greater than 7 points) in fatigue among patients with Crohn's disease taking CoQ10 to warrant conduct of a larger, placebo-controlled clinical trial. The primary outcome will be measured with the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue 7a, a unidimensional scale that has been well validated and tested among the general population and patients with IBD and many other chronic disorders. The scale ranges from 33.7 to 75.8. Higher scores indicate more greater fatigue.

SECONDARY OUTCOMES:
Change in domain specific fatigue | 8 weeks
  Secondary outcome measures will include improvement in domain specific fatigue, overall fatigue assessed with a different unidimensional scale using the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) for changes in Inflammatory Bowel Disease(IBD)-related quality of life. The scale ranges from 0 to 52. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Publication of the results of this study are planned. All publications emanating from this study will meet the authorship standards of the International Committee of Medical Journal Editors (ICMJE) standards.
  No data or samples obtained via this study will be shared with public repositories and there is no requirement to do so under the current funding mechanism for this study.
  If data or samples are shared with other investigators, they will be deidentified and the principal investigator will ensure that proper regulatory requirements are met before sharing the data. No data or samples will be provided outside of the University of Pennsylvania without an executed Material Transfer Agreement between the University of Pennsylvania and the institution receiving the data and or/samples.